CLINICAL TRIAL: NCT06725082
Title: Impact of Recombinant Humanized Type III Collagen on the Immediate and Long-term Effects of Breast Tumor Surgery: a Multicenter, Prospective, Randomized, Open-label, Parallel-controlled Trial Protocol
Brief Title: Impact of Recombinant Humanized Type III Collagen on the Immediate and Long-term Effects of Breast Tumor Surgery
Acronym: ColBreast
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shu Wang, professor，director of breast center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PKUPH2024PHD011-001
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Collagen Protein
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rhCOL3 Injection Group (Experimental): RhCOL3 will be prepared as a 4mg/ml and injected around the tumor. After the surgical margin is confirmed to be safe by rapid frozen pathology during surgery, a second injection of 2ml will be administered around the surgical area skin (at points spaced along the skin incision).
  Interventions: Biological: Recombinant Humanized Type III Collagen Injection
- Control Group (Placebo Comparator): 4ml of saline will be injected around the tumor before surgery. After the surgical margin is confirmed to be safe by rapid frozen pathology during surgery, 2ml of saline will be injected around the breast surgical area skin.
  Interventions: Biological: Recombinant Humanized Type III Collagen Injection

INTERVENTIONS:
Biological: Recombinant Humanized Type III Collagen Injection — rhCOL3/saline will be injected around the tumor (at four points: outer upper, inner upper, outer lower, and inner lower) before surgery, with 500ul per site. After the surgical margin is confirmed to be safe by rapid frozen pathology during surgery, a second injection of 2ml will be administered around the surgical area skin (at points spaced along the skin incision), followed by routine tissue flap revision and suture.

SUMMARY:
Breast tumors, particularly breast cancer, are increasingly prevalent in China, with a noticeable trend towards younger ages. Preliminary research indicates that Type III Collagen (COL3) plays a crucial role in tissue and organ protection within the tumor microenvironment and can inhibit tumor progression through microenvironmental remodeling. However, there are no clinical studies related to COL3 in breast tumors. This project aims to initiate a multicenter, prospective, randomized, open-label, parallel-controlled trial by locally administering recombinant humanized Type III Collagen (rhCOL3) to patients undergoing breast tumor surgery. The study will observe the incidence of perioperative complications after rhCOL3 injection, as well as changes in aesthetic outcomes and tumor-related pathological indicators following breast tumor surgery with local rhCOL3 injection. The goal is to establish a targeted rhCOL3 local injection therapy with dual functions of local protection and synergistic treatment, providing a new strategy for the treatment of breast tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18 years or older but not exceeding 80 years;
2. Clinical and imaging diagnosis of breast tumor, planned for needle biopsy;
3. Planned to undergo breast tumor surgery and may plan for whole-breast radiotherapy;
4. No systemic anti-tumor treatment or local treatment (including chemotherapy and radiotherapy) has been received before screening;
5. ECOG Performance Status (PS) - 0 or 1;
6. Subjects voluntarily join this study and sign the informed consent form.

Exclusion Criteria:

a.Tumor-related symptoms and treatments

1）Bilateral, multiple lesions; 2) Skin damage and ulceration on the affected side of the breast; b. History of allergy to collagen products or their excipients or severe allergic constitution; c. History of breast cancer or other malignant tumors; d. Positive serum pregnancy test or lactation; e. Use of anticoagulant drugs, such as aspirin and other non-steroidal anti-inflammatory drugs or antiplatelet drugs; f. With severe comorbidities, such as cardiovascular diseases, hematological diseases, autoimmune diseases, neurological or psychiatric disorders, etc.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Short-term postoperative complications after surgery and radiotherapy. | 3 month
  The purpose of this study is to assess the incidence rate of short-term complications within 3 months after patients complete surgery and radiotherapy. The main complications are defined as surgery or radiotherapy-related complications occurring during postoperative follow-up, including delayed wound healing, partial skin necrosis, infection, and hematoma and seroma; common adverse reactions related to breast radiotherapy include acute radiation dermatitis, breast edema, pain, etc., and late-stage breast fibrosis, edema, atrophy, telangiectasia, etc.

SECONDARY OUTCOMES:
Changes in clinical pathological indicators | 3 month
  For patients undergoing breast tumor surgery, observe changes in immune cell infiltration (CD4, CD8, FoxP3, CD80, CD206, etc.), fibroblast activation (FAP, α-SMA, S100a4, etc.), extracellular matrix remodeling (COL3A1, COL1A1), and cancer cell activation status (ki-67, P27, etc.) in postoperative pathological tissue to assess the impact of rhCOL3 on the tumor microenvironment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China, China